CLINICAL TRIAL: NCT00576420
Title: Clinical Evaluation of Efficacy and Safety of FS VH S/D 500 S-apr for Hemostasis in Subjects Undergoing Vascular Surgery
Brief Title: Fibrin Sealant Vascular Surgery Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 550602
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Results first posted 2012-11-27 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-10

CONDITIONS: Adjunct to Hemostasis in Vascular Surgery (Synthetic Vascular Grafts)
MeSH Terms: interventions — Low Density Lipoprotein Receptor-Related Protein-1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- FS VH S/D 500 s-apr - 60-Seconds (Experimental): Fibrin Sealant, Vapor Heated, Solvent/Detergent-treated with 500 IU/ml thrombin and synthetic aprotinin (FS VH S/D 500 s-apr) will be applied to the study suture line, 60-second polymerization time
  Interventions: Biological: FS VH S/D 500 s-apr, 60-seconds polymerization time
- FS VH S/D 500 s-apr - 120-Seconds (Experimental): FS VH S/D 500 s-apr will be applied to the study suture line, 120-second polymerization time
  Interventions: Biological: FS VH S/D 500 s-apr, 120-seconds polymerization time
- Control Group- Manual compression with surgical gauze pads (Active Comparator): Treatment of the study-suture line will be manual compression with surgical gauze pads.
  Interventions: Procedure: Manual compression with surgical gauze pads

INTERVENTIONS:
Biological: FS VH S/D 500 s-apr, 60-seconds polymerization time — FS VH S/D 500 s-apr (FS) is applied to the study suture line. The actual dose of FS VH S/D 500 s-apr depends on the length of the suture line and the intensity of bleeding and is to be decided by the surgeon, but the maximum dose per suture line shall not exceed 4 mL FS VH S/D 500 s apr. After application of FS VH S/D 500 s-apr to the study suture line is completed, the surgeon will wait for 1 minute to allow polymerization of FS VH S/D 500 s-apr.
  Arms: FS VH S/D 500 s-apr - 60-Seconds
Biological: FS VH S/D 500 s-apr, 120-seconds polymerization time — Treatment will be identical to the FS VH S/D 500 s-apr Group, 60 seconds polymerization time, except that the surgeons will wait 2 minutes to allow polymerization and will then open the cross clamps.
  Arms: FS VH S/D 500 s-apr - 120-Seconds
Procedure: Manual compression with surgical gauze pads — Treatment of the study suture line with manual compression with surgical gauze pads.
  Arms: Control Group- Manual compression with surgical gauze pads

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Fibrin Sealant, Vapor Heated, Solvent/Detergent-treated with 500 IU/ml thrombin and synthetic aprotinin (FS VH S/D 500 s-apr) for hemostasis in participants receiving prosthetic expanded polytetrafluoroethylene (ePTFE) conduits as compared to a control group treated by manual compression with surgical gauze pads.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of all ages
* Subject undergoing peripheral vascular surgery, ie, conduit placement with an ePTFE graft such as arterio-arterial bypasses [including: axillo-femoral, ilio-femoral, femoro-femoral, ilio-popliteal, femoro-popliteal (including below knee), femoro-tibial vessel bypass], or arteriovenous dialysis access shunt in the upper or lower extremity.
* Signed informed consent

Intraoperative inclusion criterion:

- Suture line bleeding eligible for study treatment is present after surgical hemostasis (i.e., suturing).

Suture line bleeding eligible for study treatment is defined as: any suture line bleeding that would prevent immediate closure of the wound and require treatment of the bleeding first, and on a scale of mild, moderate, and severe, the suture line bleeding is assessed as moderate or severe. (Moderate is defined as: either more than 25% of the suture line bleeds, or at least 5 suture line bleedings are present, if counting of suture line bleedings is possible, or one pulsatile suture line bleeding is present. Severe is defined as: either more than 50% of the suture line bleeds, or at least 10 suture line bleedings present, if counting of suture line bleedings is possible, or more than one pulsatile suture line bleedings are present, or at least one spurting suture line bleeding is present.)

Note: Bleedings that can be treated with additional sutures are not appropriate for the study. Such anastomoses should receive additional sutures, be re-categorized, and if they still comply with the inclusion criteria, be randomized.

Exclusion Criteria:

* Subjects concurrently participating in another clinical study treatment with another investigational drug or device within the last 30 days
* Other vascular procedures during the same surgical session (stenting and/or endarterectomy of the same artery are allowed)
* Arterio-arterial bypasses with more than 2 anastomoses (e.g., aorto-bifemoral, axillo-bifemoral etc.)
* Pregnant or lactating women
* Congenital coagulation disorders
* Prior kidney transplantation
* Heparin-induced thrombocytopenia
* Known prior exposure to aprotinin within the last 12 months
* Known hypersensitivity to aprotinin or other components of the product
* Known severe congenital or acquired immunodeficiency (e.g., HIV infection or long term treatment with immunosuppressive drugs)
* Prior radiation therapy to the operating field
* Severe local inflammation at the operating field.

Intraoperative exclusion criterion:

* Major intraoperative complications that require resuscitation or deviation from the planned surgical procedure.
* Intraoperative change in planned surgical procedure, which results in subject no longer meeting preoperative inclusion and/or exclusion criteria, (e.g. abandonment of ePTFE graft placement).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2007-12; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Birmingham, Alabama
  - Tucson, Arizona
  - Long Beach, California
  - Jacksonville, Florida
  - Lexington, Kentucky
  - Baton Rouge, Louisiana
  - Pittsburgh, Pennsylvania
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Virginia Beach, Virginia
  - Seattle, Washington

REFERENCES:
- [Result] Saha SP, Muluk S, Schenk W 3rd, Burks SG, Grigorian A, Ploder B, Presch I, Pavlova BG, Hantak E. Use of fibrin sealant as a hemostatic agent in expanded polytetrafluoroethylene graft placement surgery. Ann Vasc Surg. 2011 Aug;25(6):813-22. doi: 10.1016/j.avsg.2010.12.016. Epub 2011 Apr 21. PMID 21514114

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 12 clinical sites in the United States, beginning December 2007. The last participant completed the study in December 2008
Pre-assignment Details: 101 participants were enrolled and screened. 26 were screen failures; 1 was excluded due to study issue; and 1 was withdrawn by investigator. Therefore, 73 of the 101 enrolled were randomized and treated.
Groups:
- FS VH S/D 500 S-apr - 60 Seconds: Fibrin Sealant, Vapor Heated, Solvent/Detergent-treated with 500 IU/ml thrombin and synthetic aprotinin (FS VH S/D 500 s-apr), 60 - seconds polymerization time
- FS VH S/D 500 S-apr - 120 Seconds: FS VH S/D 500 s-apr, 120 - seconds polymerization time
- Control Group: Manual compression with surgical gauze pads.
Period: Overall Study
Arm/Group | FS VH S/D 500 S-apr - 60 Seconds | FS VH S/D 500 S-apr - 120 Seconds | Control Group
Started | 26 | 24 | 23
Completed | 26 | 24 | 22
Not Completed | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- FS VH S/D 500 S-apr - 60 Seconds: FS VH S/D 500 s-apr, 60 - seconds polymerization time
- Total: Total of all reporting groups
Arm/Group | FS VH S/D 500 S-apr - 60 Seconds | FS VH S/D 500 S-apr - 120 Seconds | Control Group | Total
Number analyzed (Participants) | 26 | 24 | 23 | 73
Age Continuous [Median (Full Range); unit: years] | 63.0 (12.7) [33 to 85] | 67.0 (14.6) [24 to 84] | 63.0 (14.4) [38 to 86] | 63 [24 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 12 | 12 | 29
  Male | 21 | 12 | 11 | 44
Region of Enrollment [Number; unit: participants]
  United States | 26 | 24 | 23 | 73

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Hemostasis at 4 Minutes After Treatment Application at the Study Suture Line.
Description: Hemostasis at the study suture line must be maintained.
  Participants were considered treatment failures if they met any of the following conditions:
  * Did not achieve hemostasis at 4 minutes
  * Required additional hemostatic treatment during the first 4 minutes of the observation period
  * Experienced rebleeding after the first 4 minutes of the observation period.
Time Frame: 4 minutes post start of treatment application
Population: Intent to Treat
Measure: Number; unit: percentage of participants
Groups:
- FS VH S/D 500 S-apr- 60-Seconds: Fibrin Sealant, Vapor Heated, Solvent/Detergent-treated with 500 IU/ml thrombin and synthetic aprotinin (FS VH S/D 500 s-apr), 60-seconds polymerization time
- FS VH S/D 500 S-apr - 120-Seconds: FS VH S/D 500 s-apr, 120-seconds polymerization time
Arm/Group | FS VH S/D 500 S-apr- 60-Seconds | FS VH S/D 500 S-apr - 120-Seconds | Control Group
Number analyzed (Participants) | 26 | 24 | 23
percentage of participants
  Primary Hemostasis Achieved at 4 Minutes | 46.2 | 62.5 | 34.8
  Additional Treatment Required for Hemostasis | 30.8 | 25.0 | 52.2
  Intraoperative Rebleeding After Primary Hemostasis | 3.8 | 0.0 | 4.3

2. Primary Outcome: 90% Confidence Interval for the Percentage of Participants Achieving Hemostasis at 4 Minutes After Treatment Application at the Suture Line
Description: Hemostasis at the study suture line must be maintained until closure of the surgical wound.
  Participants were considered treatment failures if they met any of the following conditions:
  * Did not achieve hemostasis at 4 minutes
  * Required additional hemostatic treatment other than study treatment during the first 4 minutes of the observation period
  * Experienced rebleeding after the first 4 minutes of the observation period.
Time Frame: 4 minutes post start of treatment application
Population: Intent to Treat
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- FS VH S/D 500 S-apr - 60-Seconds: FS VH S/D 500 s-apr, 60-seconds polymerization time
Arm/Group | FS VH S/D 500 S-apr - 60-Seconds | FS VH S/D 500 S-apr - 120-Seconds | Control Group
Number analyzed (Participants) | 26 | 24 | 23
percentage of participants | 46.2 [30.1 to 62.2] | 62.5 [46.2 to 78.8] | 34.8 [18.4 to 51.1]
Statistical Analysis 1: Comparison: FS VH S/D 500 S-apr - 60-Seconds vs FS VH S/D 500 S-apr - 120-Seconds vs Control Group; Test type: Superiority or Other; p = 0.1564, Likelihood ratio chi-square test

3. Primary Outcome: Hemostasis at 4 Minutes After Treatment Application at the Suture Line by Bleeding Severity - Moderate Bleeding
Description: Investigators were shown videos of bleeding severities to standardize assessments.
  1. Moderate bleeding defined as:
     * Either >25% of the suture line bleeds, or
     * ≥5 suture line bleedings were present, if counting of suture line bleedings was possible, or
     * 1 pulsatile suture line bleeding was present.
  2. Severe bleeding defined as:
     * Either >50% of the suture line bleeds, or
     * ≥10 suture line bleedings were present, if counting of suture line bleedings was possible, or
     * >1 pulsatile suture line bleeding was present, or
     * ≥1 spurting suture line bleeding was present.
Time Frame: 4 minutes post start of treatment application
Population: Intent to Treat
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | FS VH S/D 500 S-apr - 60-Seconds | FS VH S/D 500 S-apr - 120-Seconds | Control Group
Number analyzed (Participants) | 14 | 12 | 13
percentage of participants | 50.0 [28.0 to 72.0] | 66.7 [44.3 to 89.1] | 38.5 [16.3 to 60.7]

4. Secondary Outcome: Percentage of Participants Achieving Hemostasis at 6 Minutes
Description: Hemostasis at the study suture line must be maintained until closure of the surgical wound.
Time Frame: 6 minutes post start of treatment application start
Population: Intent to Treat
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | FS VH S/D 500 S-apr - 60-Seconds | FS VH S/D 500 S-apr - 120-Seconds | Control Group
Number analyzed (Participants) | 26 | 24 | 23
percentage of participants | 61.5 [45.8 to 77.2] | 75.0 [60.5 to 89.5] | 34.8 [18.4 to 51.1]
Statistical Analysis 1: Comparison: FS VH S/D 500 S-apr - 60-Seconds vs Control Group; Test type: Superiority or Other; p = 0.060, Likelihood ratio chi-square test
Statistical Analysis 2: Comparison: FS VH S/D 500 S-apr - 120-Seconds vs Control Group; Test type: Superiority or Other; p = 0.005, Likelihood ratio chi-square test

5. Secondary Outcome: Percentage of Participants Achieving Hemostasis at 10 Minutes
Description: Hemostasis at the study suture line must be maintained until closure of the surgical wound.
Time Frame: 10 minutes post start of treatment application
Population: Intent to Treat
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | FS VH S/D 500 S-apr - 60-Seconds | FS VH S/D 500 S-apr - 120-Seconds | Control Group
Number analyzed (Participants) | 26 | 24 | 23
percentage of participants | 65.4 [50.0 to 80.7] | 75.0 [60.5 to 89.5] | 43.5 [26.5 to 60.5]
Statistical Analysis 1: Comparison: FS VH S/D 500 S-apr - 60-Seconds vs Control Group; Test type: Superiority or Other; p = 0.123, Likelihood ratio chi-square test
Statistical Analysis 2: Comparison: FS VH S/D 500 S-apr - 120-Seconds vs Control Group; Test type: Superiority or Other; p = 0.026, Likelihood ratio chi-square test

6. Secondary Outcome: Percentage of Participants With Intraoperative Rebleeding After Hemostasis at the Study Suture Line
Description: Intraoperative rebleeding at the study suture line after occurrence of hemostasis.
Time Frame: Intraoperative day 0
Population: Intent to Treat
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | FS VH S/D 500 S-apr - 60-Seconds | FS VH S/D 500 S-apr - 120-Seconds | Control Group
Number analyzed (Participants) | 26 | 24 | 23
percentage of participants | 3.8 [0.0 to 10.0] | 0.0 [0.0 to 0.0] | 4.3 [0.0 to 11.3]
Statistical Analysis 1: Comparison: FS VH S/D 500 S-apr - 60-Seconds vs Control Group; Test type: Superiority or Other; p = 0.929, Likelihood ratio chi-square test
Statistical Analysis 2: Comparison: FS VH S/D 500 S-apr - 120-Seconds vs Control Group; Test type: Superiority or Other; p = 0.228, Likelihood ratio chi-square test

7. Secondary Outcome: Percentage of Participants With Postoperative Rebleeding After Hemostasis at the Study Suture Line
Description: Any rebleeding requiring surgical reexploration
Time Frame: Postoperative through day 30 ± 5
Population: Intent to Treat
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- FS VH S/D 500 S-apr - 60-Seconds: Fibrin Sealant, Vapor Heated, Solvent/Detergent-treated with 500 IU/ml thrombin and synthetic aprotinin (FS VH S/D 500 s-apr), 60-seconds polymerization time
- FS VH S/D 500 S-apr - 120-Seconds: FS VH S/D 500 s-apr, 120-seconds polymerization.
Arm/Group | FS VH S/D 500 S-apr - 60-Seconds | FS VH S/D 500 S-apr - 120-Seconds | Control Group
Number analyzed (Participants) | 26 | 24 | 23
percentage of participants | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

8. Secondary Outcome: Percentage of Participants With Any Transfusion Requirement
Description: Proportion of participants who required transfusions (i.e., red blood cell (RBC) concentrates, fresh frozen plasma (FFP), and platelets)
Time Frame: Intraoperative (day 0) through day 30 ± 5
Population: Intent to Treat
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | FS VH S/D 500 S-apr - 60-Seconds | FS VH S/D 500 S-apr - 120-Seconds | Control Group
Number analyzed (Participants) | 26 | 24 | 23
percentage of participants | 3.8 [0.0 to 10.0] | 12.5 [1.4 to 23.6] | 13.0 [1.5 to 24.6]
Statistical Analysis 1: Comparison: FS VH S/D 500 S-apr - 60-Seconds vs Control Group; Test type: Superiority or Other; p = 0.234, Likelihood ratio chi-square test
Statistical Analysis 2: Comparison: FS VH S/D 500 S-apr - 120-Seconds vs Control Group; Test type: Superiority or Other; p = 0.955, Likelihood ratio chi-square test

9. Secondary Outcome: Percentage of Participants With Graft Occlusions
Description: Determined clinically and defined as absence of blood flow through the graft.
Time Frame: Day 0 (procedure day) through day 30 ± 5
Population: Safety Analysis Set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- FS VH S/D 500 S-apr - All - (60 + 120 Seconds): All study participants who received Fibrin Sealant (60 + 120 Seconds):
  1. Fibrin Sealant, Vapor Heated, Solvent/Detergent-treated with 500 IU/ml thrombin and synthetic aprotinin (FS VH S/D 500 s-apr), 60-seconds polymerization time
  2. FS VH S/D 500 s-apr, 120-seconds polymerization time
Arm/Group | FS VH S/D 500 S-apr - 60-Seconds | FS VH S/D 500 S-apr - 120-Seconds | FS VH S/D 500 S-apr - All - (60 + 120 Seconds) | Control Group
Number analyzed (Participants) | 26 | 24 | 50 | 23
percentage of participants | 7.7 [0.0 to 16.3] | 4.2 [0.0 to 10.9] | 6.0 [0.5 to 11.5] | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: FS VH S/D 500 S-apr - 60-Seconds vs Control Group; Test type: Superiority or Other; p = 0.106, Likelihood ratio chi-square test
Statistical Analysis 2: Comparison: FS VH S/D 500 S-apr - 120-Seconds vs Control Group; Test type: Superiority or Other; p = 0.243, Likelihood ratio chi-square test
Statistical Analysis 3: Comparison: FS VH S/D 500 S-apr - All - (60 + 120 Seconds) vs Control Group; Test type: Superiority or Other; p = 0.127, Likelihood ratio chi-square test

10. Secondary Outcome: Percentage of Participants With Infections at the Surgical Site
Time Frame: Day 0 (procedure day) through day 30 ± 5
Population: Safety Analysis Set
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- FS VH S/D 500 S-apr All - (60 + 120 Seconds): All study participants who received Fibrin Sealant (60 + 120 Seconds):
  1. Fibrin Sealant, Vapor Heated, Solvent/Detergent-treated with 500 IU/ml thrombin and synthetic aprotinin (FS VH S/D 500 s-apr), 60-seconds polymerization time
  2. FS VH S/D 500 s-apr, 120-seconds polymerization time
Arm/Group | FS VH S/D 500 S-apr - 60-Seconds | FS VH S/D 500 S-apr - 120-Seconds | FS VH S/D 500 S-apr All - (60 + 120 Seconds) | Control Group
Number analyzed (Participants) | 26 | 24 | 50 | 23
percentage of participants | 3.8 [0.0 to 10.0] | 8.3 [0.0 to 17.6] | 6.0 [0.5 to 11.5] | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: FS VH S/D 500 S-apr - 60-Seconds vs Control Group; Test type: Superiority or Other; p = 0.257, Likelihood ratio chi-square test
Statistical Analysis 2: Comparison: FS VH S/D 500 S-apr - 120-Seconds vs Control Group; Test type: Superiority or Other; p = 0.096, Likelihood ratio chi-square test
Statistical Analysis 3: Comparison: FS VH S/D 500 S-apr All - (60 + 120 Seconds) vs Control Group; Test type: Superiority or Other; p = 0.127, Likelihood ratio chi-square test

11. Secondary Outcome: Vital Signs: Systolic and Diastolic Blood Pressure - Preoperative Baseline
Time Frame: Within 14 days prior to date of surgery
Population: Safety Analysis Set
Measure: Median (Full Range); unit: mm Hg
Groups:
- FS VH S/D 500 S -Apr - 60: Preoperative Baseline: FS VH S/D 500 s-apr, 60-seconds polymerization (FS 60)
- FS VH S/D 500 S -Apr - 120: Preoperative Baseline: FS VH S/D 500 s-apr, 120-seconds polymerization (FS 120)
- FS VH S/D 500 S-apr - All: Preoperative Baseline: All study participants who received Fibrin Sealant (60 + 120 Seconds polymerization time) (FS All):
  1. Fibrin Sealant, Vapor Heated, Solvent/Detergent-treated with 500 IU/ml thrombin and synthetic aprotinin (FS VH S/D 500 s-apr), 60-seconds polymerization time
  2. FS VH S/D 500 s-apr, 120-seconds polymerization time
- Control Group: Preoperative Baseline: Manual compression with surgical gauze pads
Arm/Group | FS VH S/D 500 S -Apr - 60: Preoperative Baseline | FS VH S/D 500 S -Apr - 120: Preoperative Baseline | FS VH S/D 500 S-apr - All: Preoperative Baseline | Control Group: Preoperative Baseline
Number analyzed (Participants) | 26 | 24 | 50 | 23
mm Hg
  Systolic blood pressure | 137.5 [95.0 to 182.0] | 142.5 [96.0 to 208.0] | 141.5 [95.0 to 208.0] | 150.0 [91.0 to 194.0]
  Diastolic blood pressure | 71.0 [46.0 to 100.0] | 73.5 [54.0 to 137.0] | 72.0 [46.0 to 137.0] | 78.0 [48.0 to 111.0]

12. Secondary Outcome: Percent Change in Vital Signs: Systolic and Diastolic Blood Pressure
Description: Percent Change in Systolic and Diastolic Blood Pressure (BP) Measured as: Preoperative Baseline - Intraoperative Day 0; Preoperative Baseline - Postoperative Day 1; and Preoperative Baseline - Postoperative Day 14
Time Frame: Preoperative baseline through postoperative Day 14
Population: Safety Analysis Set
Measure: Median (Full Range); unit: percent change
Groups:
- FS 60: Preoperative Baseline - Intraoperative Day 0: FS VH S/D 500 s-apr (FS), 60-seconds polymerization
- FS 120: Preoperative Baseline - Intraoperative Day 0; FS 120: Preoperative Baseline - Postoperative Day 1; FS 120: Preoperative Baseline - Postoperative Day 14: FS VH S/D 500 s-apr, 120-seconds polymerization
- FS All: Preoperative Baseline - Intraoperative Day 0; FS All: Preoperative Baseline - Postoperative Day 1; FS All: Preoperative Baseline - Postoperative Day 14: All study participants who received Fibrin Sealant (60 + 120 Seconds):
  1. Fibrin Sealant, Vapor Heated, Solvent/Detergent-treated with 500 IU/ml thrombin and synthetic aprotinin (FS VH S/D 500 s-apr), 60-seconds polymerization time
  2. FS VH S/D 500 s-apr, 120-seconds polymerization time
- Control Group: Preoperative Baseline - Intraoperative Day 0; Control Group: Preoperative Baseline - Postoperative Day 1; Control Group: Preoperative Baseline - Postoperative Day 14: Manual compression with surgical gauze pads
- FS 60: Preoperative Baseline - Postoperative Day 1; FS 60: Preoperative Baseline - Postoperative Day 14: FS VH S/D 500 s-apr, 60-seconds polymerization
Arm/Group | FS 60: Preoperative Baseline - Intraoperative Day 0 | FS 120: Preoperative Baseline - Intraoperative Day 0 | FS All: Preoperative Baseline - Intraoperative Day 0 | Control Group: Preoperative Baseline - Intraoperative Day 0 | FS 60: Preoperative Baseline - Postoperative Day 1 | FS 120: Preoperative Baseline - Postoperative Day 1 | FS All: Preoperative Baseline - Postoperative Day 1 | Control Group: Preoperative Baseline - Postoperative Day 1 | FS 60: Preoperative Baseline - Postoperative Day 14 | FS 120: Preoperative Baseline - Postoperative Day 14 | FS All: Preoperative Baseline - Postoperative Day 14 | Control Group: Preoperative Baseline - Postoperative Day 14
Number analyzed (Participants) | 26 | 24 | 50 | 23 | 26 | 24 | 50 | 23 | 25 | 22 | 47 | 20
percent change
  Systolic blood pressure | -10.1 [-36.8 to 21.4] | -6.5 [-42.2 to 44.4] | -9.8 [-42.2 to 44.4] | -17.2 [-51.5 to 15.4] | -6.4 [-34.7 to 54.1] | -12.4 [-47.1 to 62.5] | -7.9 [-47.1 to 62.5] | -11.0 [-29.5 to 44.4] | -3.8 [-29.7 to 46.9] | -3.7 [-47.1 to 50.9] | -3.8 [-47.1 to 50.9] | -6.6 [-33.5 to 10.0]
  Diastolic blood pressure | -8.2 [-66.7 to 100.0] | -16.4 [-64.6 to 36.5] | -11.4 [-66.7 to 100.0] | -21.9 [-45.0 to 41.7] | -1.5 [-38.5 to 63.0] | -19.4 [-60.6 to 40.0] | -7.5 [-60.6 to 63.0] | -9.6 [-39.4 to 13.8] | 0.0 [-28.6 to 36.7] | -7.5 [-48.9 to 51.9] | -1.1 [-48.9 to 51.9] | -7.1 [-37.5 to 39.4]

13. Secondary Outcome: Vital Signs: Heart Rate - Preoperative Baseline
Time Frame: Within 14 days prior to date of surgery
Population: Safety Analysis Set
Measure: Median (Full Range); unit: Heart beats/ minute
Groups:
- FS 60: Preoperative Baseline: FS VH S/D 500 s-apr, 60-seconds polymerization
- FS 120: Preoperative Baseline: FS VH S/D 500 s-apr, 120-seconds polymerization
- FS All: Preoperative Baseline: All study participants who received Fibrin Sealant (60 + 120 Seconds polymerization time):
  1. Fibrin Sealant, Vapor Heated, Solvent/Detergent-treated with 500 IU/ml thrombin and synthetic aprotinin (FS VH S/D 500 s-apr), 60-seconds polymerization time
  2. FS VH S/D 500 s-apr, 120-seconds polymerization time
Arm/Group | FS 60: Preoperative Baseline | FS 120: Preoperative Baseline | FS All: Preoperative Baseline | Control Group: Preoperative Baseline
Number analyzed (Participants) | 26 | 24 | 50 | 23
Heart beats/ minute | 72.0 [50.0 to 139.0] | 71.5 [53.0 to 98.0] | 72.0 [50.0 to 139.0] | 74.0 [57.0 to 112.0]

14. Secondary Outcome: Percent Change in Vital Signs: Heart Rate
Description: Percent Change in Heart Rate Measured as: Preoperative Baseline - Intraoperative Day 0; Preoperative Baseline - Postoperative Day 1; and Preoperative Baseline - Postoperative Day 14
Time Frame: Preoperative baseline through postoperative Day 14
Population: Safety Analysis Set
Measure: Median (Full Range); unit: percent change
Groups:
- FS 60: Preoperative Baseline - Intraoperative Day 0; FS 60: Preoperative Baseline - Postoperative Day 1; FS 60: Preoperative Baseline - Postoperative Day 14: FS VH S/D 500 s-apr, 60-seconds polymerization
Arm/Group | FS 60: Preoperative Baseline - Intraoperative Day 0 | FS 120: Preoperative Baseline - Intraoperative Day 0 | FS All: Preoperative Baseline - Intraoperative Day 0 | Control Group: Preoperative Baseline - Intraoperative Day 0 | FS 60: Preoperative Baseline - Postoperative Day 1 | FS 120: Preoperative Baseline - Postoperative Day 1 | FS All: Preoperative Baseline - Postoperative Day 1 | Control Group: Preoperative Baseline - Postoperative Day 1 | FS 60: Preoperative Baseline - Postoperative Day 14 | FS 120: Preoperative Baseline - Postoperative Day 14 | FS All: Preoperative Baseline - Postoperative Day 14 | Control Group: Preoperative Baseline - Postoperative Day 14
Number analyzed (Participants) | 26 | 24 | 50 | 23 | 26 | 24 | 50 | 23 | 25 | 22 | 47 | 20
percent change | -7.0 [-58.3 to 38.6] | -2.6 [-35.6 to 37.1] | -6.3 [-58.3 to 38.6] | -9.5 [-30.8 to 21.2] | -6.7 [-34.0 to 27.1] | 2.0 [-30.6 to 32.7] | -1.4 [-34.0 to 32.7] | 9.9 [-24.4 to 54.5] | 3.0 [-19.5 to 30.6] | 7.4 [-30.1 to 22.9] | 4.4 [-30.1 to 30.6] | 1.8 [-26.8 to 26.3]

15. Secondary Outcome: Vital Signs: Respiratory Rate - Preoperative Baseline
Time Frame: Within 14 days prior to date of surgery
Population: Safety Analysis Set
Measure: Median (Full Range); unit: Breaths/ minute
Arm/Group | FS 60: Preoperative Baseline | FS 120: Preoperative Baseline | FS All: Preoperative Baseline | Control Group: Preoperative Baseline
Number analyzed (Participants) | 26 | 23 | 49 | 23
Breaths/ minute | 18.0 [15.0 to 24.0] | 20.0 [13.0 to 20.0] | 18.0 [13.0 to 24.0] | 18.0 [16.0 to 26.0]

16. Secondary Outcome: Percent Change in Vital Signs: Respiratory Rate
Description: Percent Change in Respiratory Rate Measured as: Preoperative Baseline - Intraoperative Day 0; Preoperative Baseline - Postoperative Day 1; and Preoperative Baseline - Postoperative Day 14
Time Frame: Preoperative baseline through postoperative Day 14
Population: Safety Analysis Set
Measure: Median (Full Range); unit: percent change
Arm/Group | FS 60: Preoperative Baseline - Postoperative Day 1 | FS 120: Preoperative Baseline - Postoperative Day 1 | FS All: Preoperative Baseline - Postoperative Day 1 | Control Group: Preoperative Baseline - Postoperative Day 1 | FS 60: Preoperative Baseline - Postoperative Day 14 | FS 120: Preoperative Baseline - Postoperative Day 14 | FS All: Preoperative Baseline - Postoperative Day 14 | Control Group: Preoperative Baseline - Postoperative Day 14
Number analyzed (Participants) | 25 | 22 | 47 | 21 | 24 | 19 | 43 | 20
percent change | 0.0 [-35.0 to 33.3] | -10.0 [-30.0 to 28.6] | -10.0 [-35.0 to 33.3] | 0.0 [-23.1 to 25.0] | 0.0 [-20.0 to 25.0] | 0.0 [-29.4 to 38.5] | 0.0 [-29.4 to 38.5] | 0.0 [-46.2 to 33.3]

17. Secondary Outcome: Laboratory Values Over Time: Hemoglobin
Time Frame: Preoperative baseline through postoperative Day 14
Population: Safety Analysis Set
Measure: Median (Full Range); unit: g/dl
Groups:
- FS All: Preoperative Baseline; FS All: Postoperative Day 14: All study participants who received Fibrin Sealant (60 + 120 Seconds):
  1. Fibrin Sealant, Vapor Heated, Solvent/Detergent-treated with 500 IU/ml thrombin and synthetic aprotinin (FS VH S/D 500 s-apr), 60-seconds polymerization time
  2. FS VH S/D 500 s-apr, 120-seconds polymerization time
- FS 60: Postoperative Day 14: FS VH S/D 500 s-apr, 60-seconds polymerization
- FS 120: Postoperative Day 14: FS VH S/D 500 s-apr, 120-seconds polymerization
- Control Group: Postoperative Day 14: Manual compression with surgical gauze pads
Arm/Group | FS 60: Preoperative Baseline | FS 120: Preoperative Baseline | FS All: Preoperative Baseline | Control Group: Preoperative Baseline | FS 60: Postoperative Day 14 | FS 120: Postoperative Day 14 | FS All: Postoperative Day 14 | Control Group: Postoperative Day 14
Number analyzed (Participants) | 24 | 22 | 46 | 20 | 26 | 20 | 46 | 18
g/dl | 12.00 [6.60 to 16.50] | 12.55 [9.00 to 16.60] | 12.25 [6.60 to 16.60] | 12.15 [10.10 to 14.70] | 11.15 [7.60 to 16.10] | 12.40 [8.30 to 14.40] | 12.05 [7.60 to 16.10] | 11.70 [8.50 to 13.60]

18. Secondary Outcome: Laboratory Values Over Time: Hematocrit
Time Frame: Preoperative baseline through postoperative Day 14
Population: Safety Analysis Set
Measure: Median (Full Range); unit: percentage of red blood cells in blood
Arm/Group | FS 60: Preoperative Baseline | FS 120: Preoperative Baseline | FS All: Preoperative Baseline | Control Group: Preoperative Baseline | FS 60: Postoperative Day 14 | FS 120: Postoperative Day 14 | FS All: Postoperative Day 14 | Control Group: Postoperative Day 14
Number analyzed (Participants) | 24 | 22 | 46 | 20 | 26 | 20 | 46 | 18
percentage of red blood cells in blood | 37.00 [23.00 to 47.00] | 37.00 [30.00 to 51.00] | 37.00 [23.00 to 51.00] | 39.00 [30.00 to 45.00] | 35.00 [26.00 to 48.00] | 38.00 [28.00 to 47.00] | 37.00 [26.00 to 48.00] | 36.50 [27.00 to 41.00]

19. Secondary Outcome: Laboratory Values Over Time: Erythrocytes
Time Frame: Preoperative baseline through postoperative Day 14
Population: Safety Analysis Set
Measure: Median (Full Range); unit: x10^6/µl
Arm/Group | FS 60: Preoperative Baseline | FS 120: Preoperative Baseline | FS All: Preoperative Baseline | Control Group: Preoperative Baseline | FS 60: Postoperative Day 14 | FS 120: Postoperative Day 14 | FS All: Postoperative Day 14 | Control Group: Postoperative Day 14
Number analyzed (Participants) | 24 | 22 | 46 | 20 | 26 | 20 | 46 | 18
x10^6/µl | 4.10 [3.10 to 5.30] | 4.15 [3.10 to 5.30] | 4.10 [3.10 to 5.30] | 4.40 [3.30 to 5.00] | 3.75 [2.90 to 5.40] | 4.15 [2.80 to 5.80] | 3.90 [2.80 to 5.80] | 4.00 [2.90 to 4.70]

20. Secondary Outcome: Laboratory Values Over Time: Leukocytes, Basophils, Eosinophils, Lymphocytes, Neutrophils, and Monocytes
Time Frame: Preoperative baseline through postoperative Day 14
Population: Safety Analysis Set
Measure: Median (Full Range); unit: x10^3/µl
Arm/Group | FS 60: Preoperative Baseline | FS 120: Preoperative Baseline | FS All: Preoperative Baseline | Control Group: Preoperative Baseline | FS 60: Postoperative Day 14 | FS 120: Postoperative Day 14 | FS All: Postoperative Day 14 | Control Group: Postoperative Day 14
Number analyzed (Participants) | 24 | 22 | 46 | 20 | 26 | 20 | 46 | 18
x10^3/µl
  Leukocytes | 6.31 [2.48 to 16.22] | 7.14 [3.45 to 15.16] | 6.62 [2.48 to 16.22] | 7.98 [3.62 to 13.76] | 6.58 [3.34 to 14.12] | 7.87 [4.36 to 16.89] | 7.00 [3.34 to 16.89] | 8.13 [6.25 to 18.62]
  Basophils | 0.05 [0.00 to 0.12] | 0.05 [0.00 to 0.10] | 0.05 [0.00 to 0.12] | 0.04 [0.00 to 0.10] | 0.04 [0.00 to 0.19] | 0.05 [0.02 to 0.23] | 0.05 [0.00 to 0.23] | 0.04 [0.00 to 0.08]
  Eosinophils | 0.17 [0.02 to 0.91] | 0.14 [0.02 to 0.96] | 0.15 [0.02 to 0.96] | 0.19 [0.04 to 0.83] | 0.21 [0.02 to 0.96] | 0.24 [0.01 to 0.52] | 0.23 [0.01 to 0.96] | 0.21 [0.08 to 0.46]
  Lymphocytes | 1.50 [0.57 to 3.86] | 1.74 [0.56 to 3.10] | 1.55 [0.56 to 3.86] | 1.59 [1.09 to 4.26] | 1.50 [0.60 to 4.59] | 1.46 [0.51 to 3.11] | 1.48 [0.51 to 4.59] | 1.94 [0.86 to 3.82]
  Neutrophils | 3.70 [1.59 to 12.55] | 4.69 [2.22 to 13.70] | 4.11 [1.59 to 13.70] | 5.24 [2.17 to 8.67] | 4.44 [2.38 to 9.92] | 5.23 [2.72 to 15.38] | 4.66 [2.38 to 15.38] | 5.54 [3.81 to 14.64]
  Monocytes | 0.34 [0.08 to 0.72] | 0.41 [0.20 to 0.82] | 0.36 [0.08 to 0.82] | 0.39 [0.18 to 0.83] | 0.35 [0.22 to 0.58] | 0.43 [0.22 to 0.77] | 0.38 [0.22 to 0.77] | 0.44 [0.13 to 0.57]

21. Secondary Outcome: Laboratory Values Over Time: Platelets
Time Frame: Preoperative baseline through postoperative Day 14
Population: Safety Analysis Set
Measure: Median (Full Range); unit: x10^3/µl
Arm/Group | FS 60: Preoperative Baseline | FS 120: Preoperative Baseline | FS All: Preoperative Baseline | Control Group: Preoperative Baseline | FS 60: Postoperative Day 14 | FS 120: Postoperative Day 14 | FS All: Postoperative Day 14 | Control Group: Postoperative Day 14
Number analyzed (Participants) | 23 | 19 | 42 | 19 | 25 | 19 | 44 | 16
x10^3/µl | 184.00 [70.00 to 423.00] | 204.00 [56.00 to 442.00] | 195.50 [56.00 to 442.00] | 233.00 [132.00 to 462.00] | 226.00 [138.00 to 538.00] | 333.00 [117.00 to 593.00] | 275.00 [117.00 to 593.00] | 295.00 [199.00 to 386.00]

22. Secondary Outcome: Laboratory Values Over Time: Creatinine, Bilirubin, and Blood Urea Nitrogen (BUN)
Time Frame: Preoperative baseline through postoperative Day 14
Population: Safety Analysis Set
Measure: Median (Full Range); unit: mg/dL
Arm/Group | FS 60: Preoperative Baseline | FS 120: Preoperative Baseline | FS All: Preoperative Baseline | Control Group: Preoperative Baseline | FS 60: Postoperative Day 14 | FS 120: Postoperative Day 14 | FS All: Postoperative Day 14 | Control Group: Postoperative Day 14
Number analyzed (Participants) | 25 | 24 | 49 | 20 | 26 | 21 | 47 | 18
mg/dL
  Creatinine | 4.20 [0.50 to 13.80] | 1.90 [0.60 to 13.30] | 3.50 [0.50 to 13.80] | 2.65 [0.50 to 9.40] | 4.60 [0.60 to 12.70] | 2.40 [0.60 to 12.70] | 3.50 [0.60 to 12.70] | 3.25 [0.50 to 11.00]
  Bilirubin | 0.40 [0.20 to 1.00] | 0.30 [0.20 to 1.10] | 0.30 [0.20 to 1.10] | 0.40 [0.20 to 0.70] | 0.30 [0.20 to 3.30] | 0.40 [0.20 to 0.70] | 0.30 [0.20 to 3.30] | 0.30 [0.20 to 0.60]
  BUN | 24.00 [6.00 to 104.00] | 31.00 [8.00 to 122.00] | 26.00 [6.00 to 122.00] | 29.00 [9.00 to 73.00] | 30.00 [4.00 to 72.00] | 26.00 [8.00 to 125.00] | 27.00 [4.00 to 125.00] | 27.00 [6.00 to 84.00]

23. Secondary Outcome: Laboratory Values Over Time: Alanine Aminotransferase (ALT)
Time Frame: Preoperative baseline through postoperative Day 14
Population: Safety Analysis Set
Measure: Median (Full Range); unit: U/L
Arm/Group | FS 60: Preoperative Baseline | FS 120: Preoperative Baseline | FS All: Preoperative Baseline | Control Group: Preoperative Baseline | FS 60: Postoperative Day 14 | FS 120: Postoperative Day 14 | FS All: Postoperative Day 14 | Control Group: Postoperative Day 14
Number analyzed (Participants) | 25 | 23 | 48 | 20 | 26 | 21 | 47 | 18
U/L | 16.00 [4.00 to 47.00] | 17.00 [7.00 to 43.00] | 16.00 [4.00 to 47.00] | 16.50 [7.00 to 29.00] | 12.00 [4.00 to 32.00] | 15.00 [4.00 to 39.00] | 14.00 [4.00 to 39.00] | 12.00 [4.00 to 20.00]

24. Secondary Outcome: Laboratory Values Over Time: Aspartate Aminotransferase (AST)
Time Frame: Preoperative baseline through postoperative Day 14
Population: Safety Analysis Set
Measure: Median (Full Range); unit: U/L
Arm/Group | FS 60: Preoperative Baseline | FS 120: Preoperative Baseline | FS All: Preoperative Baseline | Control Group: Preoperative Baseline | FS 60: Postoperative Day 14 | FS 120: Postoperative Day 14 | FS All: Postoperative Day 14 | Control Group: Postoperative Day 14
Number analyzed (Participants) | 25 | 22 | 47 | 19 | 26 | 19 | 45 | 18
U/L | 18.00 [14.00 to 51.00] | 19.00 [11.00 to 45.00] | 18.00 [11.00 to 51.00] | 16.00 [12.00 to 44.00] | 18.00 [13.00 to 29.00] | 20.00 [7.00 to 39.00] | 19.00 [7.00 to 39.00] | 17.50 [11.00 to 30.00]

25. Secondary Outcome: Laboratory Values Over Time: Activated Partial Thromboplastin Time (aPTT)
Time Frame: Preoperative baseline through postoperative Day 14
Population: Safety Analysis Set
Measure: Median (Full Range); unit: seconds
Arm/Group | FS 60: Preoperative Baseline | FS 120: Preoperative Baseline | FS All: Preoperative Baseline | Control Group: Preoperative Baseline | FS 60: Postoperative Day 14 | FS 120: Postoperative Day 14 | FS All: Postoperative Day 14 | Control Group: Postoperative Day 14
Number analyzed (Participants) | 22 | 21 | 43 | 20 | 24 | 18 | 42 | 18
seconds | 25.10 [19.60 to 109.80] | 26.30 [21.60 to 51.00] | 25.90 [19.60 to 109.80] | 25.10 [19.90 to 150.00] | 24.65 [20.30 to 150.00] | 27.20 [20.10 to 150.00] | 25.00 [20.10 to 150.00] | 26.75 [20.40 to 150.00]

26. Secondary Outcome: Laboratory Values Over Time: International Normalized Ratio (INR)
Time Frame: Preoperative baseline through postoperative Day 14
Population: Safety Analysis Set
Measure: Median (Full Range); unit: ratio
Arm/Group | FS 60: Preoperative Baseline | FS 120: Preoperative Baseline | FS All: Preoperative Baseline | Control Group: Preoperative Baseline | FS 60: Postoperative Day 14 | FS 120: Postoperative Day 14 | FS All: Postoperative Day 14 | Control Group: Postoperative Day 14
Number analyzed (Participants) | 21 | 21 | 42 | 20 | 24 | 17 | 41 | 18
ratio | 1.00 [0.90 to 1.20] | 1.10 [1.00 to 2.40] | 1.00 [0.90 to 2.40] | 1.05 [0.90 to 1.20] | 1.00 [0.90 to 2.10] | 1.00 [0.90 to 3.20] | 1.00 [0.90 to 3.20] | 1.00 [0.90 to 4.10]

27. Primary Outcome: Hemostasis at 4 Minutes After Treatment Application at the Suture Line by Bleeding Severity - Severe Bleeding
Description: Investigators were shown videos of bleeding severities to standardize assessments.
  Severe bleeding defined as:
  * Either >50% of the suture line bleeds, or
  * ≥10 suture line bleedings were present, if counting of suture line bleedings was possible, or
  * >1 pulsatile suture line bleeding was present, or
  * ≥1 spurting suture line bleeding was present.
Time Frame: 4 minutes post start of treatment application
Population: Intent to Treat
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | FS VH S/D 500 S-apr - 60-Seconds | FS VH S/D 500 S-apr - 120-Seconds | Control Group
Number analyzed (Participants) | 12 | 12 | 10
percentage of participants | 41.7 [18.3 to 65.1] | 58.3 [34.9 to 81.7] | 30.0 [6.2 to 53.8]

ADVERSE EVENTS:
Time Frame: Throughout study period (1 year)
Groups:
- Fibrin Sealant - 60 Seconds: Fibrin Sealant, Vapor Heated, Solvent/Detergent-treated with 500 IU/ml thrombin and synthetic aprotinin (FS VH S/D 500 s-apr), 60 seconds polymerization time
- Fibrin Sealant - 120 Seconds: FS VH S/D 500 s-apr, 120 seconds polymerization time
- Fibrin Sealant All - (60 + 120 Seconds): All study participants who received Fibrin Sealant (60 + 120 Seconds):
  1. Fibrin Sealant, Vapor Heated, Solvent/Detergent-treated with 500 IU/ml thrombin and synthetic aprotinin (FS VH S/D 500 s-apr), 60 seconds polymerization time
  2. FS VH S/D 500 s-apr, 120 seconds polymerization time
- Control Group: Treatment of the study-suture line will be manual compression with surgical gauze pads.
Arm/Group | Fibrin Sealant - 60 Seconds | Fibrin Sealant - 120 Seconds | Fibrin Sealant All - (60 + 120 Seconds) | Control Group
Serious Adverse Events (participants affected / at risk) | 4/26 | 4/24 | 8/50 | 4/23
Other Adverse Events (participants affected / at risk) | 4/26 | 9/24 | 13/50 | 7/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fibrin Sealant - 60 Seconds (N=26) | Fibrin Sealant - 120 Seconds (N=24) | Fibrin Sealant All - (60 + 120 Seconds) (N=50) | Control Group (N=23)
Graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Incision site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vascular graft complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fibrin Sealant - 60 Seconds (N=26) | Fibrin Sealant - 120 Seconds (N=24) | Fibrin Sealant All - (60 + 120 Seconds) (N=50) | Control Group (N=23)
Incision site complication (Injury, poisoning and procedural complications) | 2 (3) | 2 (2) | 4 (5) | 0 (0)
Incision site oedema (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Incision site erythema (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Ventricular tachycardia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxter's agreements with PIs may vary per requirements of the individual PI, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication or 1 year after study completion. Baxter requires a review of results communications (e.g., for confidential information) ≥45 days prior to submission or communication. Baxter may request an additional delay of ≤60 days (e.g., for intellectual property protection)